CLINICAL TRIAL: NCT02477072
Title: A Pilot Study on the Influence of an Optimized Heparin Regimen on the Hemostatic Environment Downstream From the Surgical Clamp in Major Vascular Surgery.
Brief Title: Optimized Heparin Regimen in Vascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15.077
Record Dates: First submitted 2015-06-16; First posted 2015-06-22 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Peripheral Revascularisation
MeSH Terms: interventions — Thrombelastography; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed heparin dose (general anesthesia) (Active Comparator): Study subjects will be randomized to receive a fixed dose of 5000 units of heparin administered intravenously 2 minutes prior to vascular clamping and blood flow interruption. A subsequent dose of heparin will be administered if requested by the surgeon following a visual assessment of the anticoagulation in the surgical field. Anticoagulation will be monitored at different time points during surgery using ACT and TEG. Peripheral blood flow will be assessed prior and after surgery using the ankle-brachial index and toe-brachial index.
  Interventions: Procedure: ACT; Procedure: TEG; Procedure: Ankle-brachial index; Procedure: Toe-brachial index; Drug: Heparin
- Weight-adjusted doses of heparin (Experimental): Study subjects will be randomized to receive 100 units of heparin per kilogram administered intravenously 2 minutes before vascular clamping and blood flow interruption. Subsequent doses of heparin will be administered to maintain the ACT between 300 and 350 seconds at all times during vascular clamping. Anticoagulation will be monitored at different time points during surgery using ACT and TEG. Peripheral blood flow will be assessed prior and after surgery using the ankle-brachial index and toe-brachial index.
  Interventions: Procedure: ACT; Procedure: TEG; Procedure: Ankle-brachial index; Procedure: Toe-brachial index; Drug: Heparin
- Fixed heparin dose (regional anesthesia) (Active Comparator): For safety reasons, study subjects under regional anesthesia will automatically be assigned to this group and will receive a fixed dose of 5000 units of heparin administered intravenously 2 minutes prior to vascular clamping and blood flow interruption. A subsequent dose of heparin will be administered if requested by the surgeon following a visual assessment of the anticoagulation in the surgical field. Anticoagulation will be monitored at different time points during surgery using ACT and TEG.
  Interventions: Procedure: ACT; Procedure: TEG; Drug: Heparin

INTERVENTIONS:
Procedure: ACT — Blood samples for ACT will be collected following induction of anesthesia, 30 minutes after heparin administration, and on arrival in the recovery room.
  Other Names: Activated clotting time
Procedure: TEG — Blood samples for TEG will be collected following induction of anesthesia, 30 minutes after heparin administration, and on arrival in the recovery room.
  Other Names: Thromboelastography
Procedure: Ankle-brachial index — Peripheral blood flow will be assessed prior and after surgery using the ankle-brachial and toe-brachial indexes.
  Arms: Fixed heparin dose (general anesthesia); Weight-adjusted doses of heparin
Procedure: Toe-brachial index — Peripheral blood flow will be assessed prior and after surgery using the ankle-brachial and toe-brachial indexes.
  Arms: Fixed heparin dose (general anesthesia); Weight-adjusted doses of heparin
Drug: Heparin — Heparin doses will be administered according to the assigned group.
  Other Names: Unfractionated heparin

SUMMARY:
Hypothesis: Optimal anticoagulation defined as an Activated Clotting Time (ACT) of 300 to 350 seconds obtained by weight-adjusted doses of unfractionated heparin (UFH) will improve the hemostatic environment downstream from the vascular clamp, provide better blood flow in the distal bed following peripheral revascularization surgery.

Objectives: This study is designed to assess the effects of an optimized regimen of UFH on the hemostatic environment downstream from the vascular clamp in major vascular surgery.

DETAILED DESCRIPTION:
Peripheral revascularization surgery is usually performed in high-risk patients, suffering from major comorbidities. Complications associated with vascular surgery include coronary problems, arrhythmias, failure of revascularization and thrombosis. In order to prevent these complications and possible re-interventions it is essential to optimize the intraoperative path.

Unfractionated heparin is commonly used during arterial vascular surgery to prevent thrombosis and accumulation of thrombi at the surgical site. UFH is administered before clamping and blood flow interruption. However, the best heparin regimen to achieve optimal anticoagulation for peripheral revascularization remains unknown, with current recommendations based on data from the coronary literature and guidelines. Few studies have assessed the effect of vascular clamping and blood flow interruption on the anticoagulation in the distal vascular bed.

Perioperative monitoring of coagulation is important to diagnose potential causes of hemorrhage and guide hemostatic therapies. Routine laboratory-based coagulation tests such as prothrombin time (PT), International Normalized Ratio (INR), activated partial thromboplastin time (aPTT) and platelet count are used to assess the patient's coagulation status. However, the value of these tests has been questioned in the acute perioperative setting for the following reasons: substantial delays between blood sampling and results, tests performed on plasma rather than whole blood and lack of information on platelet function.

The activated clotting time (ACT) is used to monitor anticoagulation and, indirectly, concentrations of UFH. The ACT is measured on whole blood in cuvettes containing high concentrations of activators, typically celite or kaolin. Modern methods are completely automated. ACT measurement with point-of-care devices is used during procedures requiring anticoagulation, such as cardiopulmonary bypass, interventional cardiology and hemodialysis. In vascular surgery, the target ACT is not clearly defined and therefore not systematically monitored.

Thromboelastography (TEG) is a bedside coagulation test that enables evaluation of all components of hemostasis. An advantage of TEG over conventional tests of hemostasis is that it is performed on whole blood, taking into consideration the role of interacting blood elements. The TEG can also be adapted to different clinical situations. Activators such as tissue factor, celite and thrombin can be added to whole blood to accelerate the analysis. TEG cups coated with heparinase can also be used to degrade heparin without affecting other coagulation parameters.

Ankle-brachial (ABI) and toe-brachial (TBI) indexes are currently used to evaluate patients with peripheral arterial disease. These non-invasive tests provide information about peripheral blood flow. The ankle-brachial index is the ratio of the systolic blood pressure at the ankle to that measured at the brachial artery. The diagnostic limits of the ABI have been confirmed in several large-scale studies. Conditions associated with medial calcifications, such as diabetes, chronic kidney disease or advanced age, can lead to false results due to vessel stiffness. The toe vessels are less susceptible to vessel stiffness, which makes the TBI useful.

Methods:

Monitoring and postoperative analgesia will be left to the discretion of the attending anesthesiologist. Surgery will be performed under general or regional anesthesia. For safety reasons, patients under regional anesthesia will automatically be assigned to receive a fixed dose of heparin.

UFH will be administered 2 minutes prior to vascular clamping according to randomization. Blood samples will be collected at the following time points for ACT and TEG analysis: following induction of anesthesia, 30 minutes after heparin administration, and on arrival in the recovery room. Heparin will be neutralized with protamine if needed.

Intraoperative blood losses will be recorded. Administration of crystalloids, colloids and blood products during surgery will be noted. Blood samples to assess cardiac troponin levels will be collected in the recovery room and on the day following surgery. Ankle-brachial and toe-brachial indexes will be measured preoperatively and postoperatively in the recovery room. The occurrence of cardiovascular complications will be noted during the hospital stay. The incidence of vascular re-interventions will be noted 30 days following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective revascularization surgery
* American Society of Anesthesiologists (ASA) physical status l-lll inclusive

Exclusion Criteria:

* Known or suspected allergy to heparin or protamine
* Contraindication to heparin or protamine
* Known or suspected coagulopathy
* Current anticoagulation or residual effect of anticoagulants, antiplatelet agents, except aspirin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Anticoagulation upstream and downstream from the clamp | From induction of anesthesia until 30 minutes following the return of normal blood flow
  Adequacy of anticoagulation upstream and downstream from the clamp will be assessed with the ACT and the thromboelastogram.

SECONDARY OUTCOMES:
Peripheral blood flow | Before surgery and following surgery in the recovery room - on Day 1
  Peripheral blood flow will be assessed by the toe-brachial and ankle-brachial indexes
Occurence of any new revascularization surgery as a measure of safety and efficacy | From surgery until thirty days following surgery
Occurrence of arrhythmia as a measure of safety | From surgery until discharge from the hospital - approximately 4 days
Quantity of blood lost during surgery as a measure of safety | At the end of surgery - on Day 1
Number of red blood cells transfusions administered as a measure of safety | From surgery until discharge from the hospital - approximately 4 days
Occurence of thrombosis as a measure of safety | From surgery until discharge from the hospital - approximately 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Hardy Jean-François, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM-Hôtel-Dieu), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Roy M, Todorov A, Ruel M, Elkouri S, Hardy JF. Anticoagulation Obtained below the Arterial Clamp Using a Single Fixed Bolus of Heparin in Vascular Surgery: A Pilot Study. Ann Vasc Surg. 2018 Jul;50:242-248. doi: 10.1016/j.avsg.2017.11.060. Epub 2018 Feb 23. PMID 29481926